CLINICAL TRIAL: NCT05486104
Title: A Multicenter, Randomized, Double-blind, Placebo Parallel Controlled Clinical Study on the Effecacy and Safety of Low-High Dosing Regimens of Hemay005 in Patients With Moderate to Severe Ulcerative Colitis
Brief Title: Phase II Study of Hemay005 in Patients With Active Ulcerative Colitis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ganzhou Hemay Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HM005UC2S01
Record Dates: First submitted 2022-08-01; First posted 2022-08-03 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Moderate to Severe Ulcerative Colitis
MeSH Terms: interventions — Hemay005

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Hemay005 45 mg BID group (Experimental): 3 tablets of Hemay005 (15mg/tablet) and 1 tablet of Hemay005 placebo will be orally administered twice daily.
  Interventions: Drug: Hemay005 tablets; Drug: Hemay005 placebo tablets
- Hemay005 60 mg BID group (Experimental): 4 tablets of Hemay005 (15mg/tablet) will be orally administered twice daily.
  Interventions: Drug: Hemay005 tablets
- Hemay005 placebo BID group (Placebo Comparator): 4 tablets of Hemay005 placebo will be orally administered twice daily.
  Interventions: Drug: Hemay005 placebo tablets

INTERVENTIONS:
Drug: Hemay005 tablets — Hemay005 tablets (15mg/tablet）will be orally administered twice daily.
  Other Names: Hemay005 45 mg BID group
  Arms: Hemay005 45 mg BID group; Hemay005 60 mg BID group
Drug: Hemay005 placebo tablets — Hemay005 placebo tablets will be orally administered twice daily.
  Other Names: Hemay005 placebo BID group
  Arms: Hemay005 45 mg BID group; Hemay005 placebo BID group

SUMMARY:
This study is a multicenter, randomized, double-blind study. There are three dosage groups: Hemay005 45 mg BID group, 60 mg BID group or placebo group, with 36 patients in each dosage group. All patients will enter a 12-week double-blind treatment period. All subjects who have received the investigational drug should be subjected to a 4-week observation after the end of treatment.

DETAILED DESCRIPTION:
This study adopts a multicenter, randomized, double-blind, low--high dose groups and placebo parallel controlled clinical study design. After screening, patients with active ulcerative colitis who meet the inclusion criteria and do not meet the exclusion criteria will be randomized by 1:1:1 to Hemay005 45 mg BID group, 60 mg BID group or placebo group, with proposed 36 patients in each group. All patients will enter a 12-week double-blind inductive treatment period. All randomized subjects who have received the investigational drug should be subjected to a 4-week observation after the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in the trial and signing the informed consent forms;
* Age ≥18 years old, male or female;
* Diagnosed as ulcerative colitis (UC) ≥ 3 months at screening with clinical manifestations and evidence of endoscopy and confirmed by histopathological reports;
* Expansion of the affected bowel segment beyond the rectum confirmed on endoscopy (affected bowel segment≥15cm);
* Moderate to severe ulcerative colitis with Modified Mayo clinical score (MMCS)≥ 4 points and ≤9 points, the Endoscopy subscore ≥ 2 points within 14 days before randomization and Stool Frequency subscore ≥ 1 point;
* UC treatment failure or intolerance (intolerance is defined as the discontinuation of drug use due to adverse reactions judged by the investigators) experienced by patients using at least one of the following:

Oral administration of sulfasalazine (SASP) and/or 5-aminosalicylic acid (5-ASA); Oral administration of corticosteroids; Azathioprine or 6-mercaptopurine; Anti-TNF-α treatment: infliximab or adalimumab, etc.; - If the patient is using the following drugs to treat ulcerative colitis at the time of screening, it is necessary to receive stable treatment during the screening period and the following requirements during the study period are as follows: Oral administration of sulfasalazine (SASP) and/or 5-aminosalicylic acid (5-ASA) maintaining stable for at least ≥ 2 weeks prior to endoscopy during the screening period and maintaining stable during the study period; and/or Oral administration of low-dose corticosteroids (≤25 mg/d prednisolone or equivalent drug dose) maintaining stable for at least ≥ 2 weeks prior to endoscopy during the screening period;

- At least one of the following effective contraceptive methods should be adopted for female patients with fertility and male patients who have not undergone vasectomy during the entire study period from the date of signing the informed consent to 3 months after the last dose. Acceptable contraceptive methods in this study include: a. abstinence; b. hormones (oral intake, patch, ring, injection, implantation) combined with male condoms. This measure must be applied at least 30 days prior to the first administration of investigational drug, otherwise another acceptable method of contraception must be used; c. intra-uterine device (IUD) combined with male condoms; d. barrier method (diaphragm, cervical cap, sponge) combined with male condoms; exceptional circumstances: a) females who have been menopausal for 5 years and more, and b) surgical sterilization (proof should be provided).

Exclusion Criteria:

* Pregnant or lactating women, or women or men whose partners planning to become pregnant during the study;
* Knownto be allergic to any component of Hemay005 tablets (the main component is hemay005, and the main excipients are mannitol, low substituted hydroxypropyl cellulose, croscarmellose sodium and magnesium stearate);
* Patients with suspected or confirmed Crohn's disease, undiagnosed types of colitis, fulminant colitis, toxic megacolon, microscopic colitis, ischemic colitis or radioactive colitis based on medical history and endoscopy and/or histological results;
* Patients with active EBV and/or CMV infection (EBV antibody IgM and/or EBV DNA positive); CMV antibody IgM and/or CMV DNA positive);
* Patients with the disease confined to the rectum (ulcerative proctitis) according to the endoscopy during screening;
* Patients who have undergone surgical treatment for ulcerative colitis or who require surgery during the study;
* Patients with active infection or positive pathogen test at the time of screening, and determined by the investigator to increase the risk of the subject, except for those with negative repeat test results and no symptoms of persistent infection (if time permits, during screening treatment and repeat testing);
* Patients receiving the following treatments:

Patients who have used azathioprine/6-mercaptopurine, methotrexate within 7 days before randomization; Patients who have used cyclosporine, mycophenolate mofetil, tacrolimus/sirolimus within 4 weeks before randomization; Patients who have used interferon within 8 weeks before randomization; Patients who have received anti-TNF-α treatment within 8 weeks before randomization; Intravenous corticosteroids or rectal administration of corticosteroids or rectal administration of 5-ASA within 2 weeks prior to randomization; Patients who have used thalidomide within 8 weeks before randomization;Patients who have received antibiotic treatment within 1 week before randomization;

* Patients with active infection and judged by the investigator to increase the risk of the subjects;
* Patients with a history of TB or active TB (Investigator-judged signs or symptoms of active tuberculosis at screening):

Screening was permitted if patients had a history of tuberculosis and had been cured by investigator assessment for at least 3 years prior to randomization; subjects with a negative T-cell test for tuberculosis infection (T-SPOT) at screening can be included in this study. Subjects who are T-SPOT positive during the screening period need to undergo tuberculosis-related clinical examinations (Tuberculosis-related clinical work performed within 12 weeks prior to randomization can be used directly for evaluation), if the tuberculosis-related clinical examination confirmed active tuberculosis, the subjects will not be eligible for this study. Subjects can be included in this study if the tuberculosis-related clinical examination confirms inactive tuberculosis. If the research center cannot perform T-SPOT test, TB screening by QuantiFERON-TB Gold test kit can also be accepted. The treatment of QuantiFERON-TB-Gold screening results is the same as that of T-SPOT.

* Patients with hemoglobin <8 g/dL or hematocrit <30%, white blood cells <3.0 × 10^9/L or neutrophils <1.2 × 10^9/L, platelets <100 × 10^09/L at screening;
* Total bilirubin (TBIL), aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥ 2 upper limits of normal (ULN) at screening;
* Glomerular filtration rate (eGFR) ≤ 40 ml/min;
* Patients with hereditary immunodeficiency disease;
* Patients with a history of lymphoproliferative disorders (e.g. EBV-related lymphoproliferative disorders), or with lymphoma, leukemia, myeloproliferative disease, multiple myeloma;
* Lymphocyte apheresis or selective mononuclear granulocyte apheresis was performed within 12 months before the screening or is planned to be performed during the study;
* Patients with malignant tumor or with a history of malignancy other than well-treated or resected basal cell or squamous cell skin cancer;
* Patients with conditions that may affect oral drug absorption, e.g. gastrectomy or clinically significant diabetes-related gastrointestinal disorders, or specific types of obesity surgery such as gastric bypass, however, patients only subjected to the division of the stomach into independent chambers, like gastric banding, will not be excluded;
* Patients with previous surgery on small intestine or colon and with evidence of colonic dysplasia or intestinal stenosis;
* Patients with chronic hepatitis B virus (HBV) infection (hepatitis B surface antigen (HBsAg), hepatitis B surface antibody (HBsAb) and hepatitis B core antibody (HBcAb) should be assessed for all patients during screening: patients with positive hepatitis B surface antigen (HBsAg) will be excluded; patients with HBsAg (negative), HBsAb (negative or positive) and HBcAb (positive) should be tested for HBV-DNA, and if the HBV-DNA result is positive, patient will be excluded; if the HBV-DNA result is negative, patients can be enrolled in the study.), chronic hepatitis C virus (HCV) infection (patients with positive hepatitis C virus antibody (HCVAb) excluded) or human immunodeficiency virus (HIV) infection (patients with positive human immunodeficiency virus (HIV) antibody excluded) or Syphilis (TP) infection (excluded patients with Treponema pallidum antibody (Anti-TP) positive);
* Patients receive any live vaccine at present or has received any live vaccine within 8 weeks prior to randomization, or have been vaccinated against COVID-19 within 14 days prior to randomization;
* Use of cytochrome P450 enzyme inducers (such as rifampicin, phenobarbital, dexamethasone, isoniazid, carbamazepine, etc.) within 14 days before screening;
* Suicidal behavior (including active attempts, interrupted attempts, or attempted attempts) or suicidal thoughts within the past 6 months;
* Other conditions that the investigator judges as unsuitable to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
clinical remission | 12 week
  Definition of clinical remission rate: defined as a Mayo score of 0 or 1 in the number of bowel movements with a ≥1 reduction from baseline, a blood in the stool score of 0, and an endoscopic score of 0 or 1 (no fragility).

SECONDARY OUTCOMES:
clinical response | 12 week
  Definition of clinical response: defined as a Mayo score reduction of ≥2 points from baseline and a decrease of ≥30% from baseline, with a reduction of ≥1 point from baseline in the rectal bleeding sub-score, or a rectal bleeding sub-score of ≤1 point.

CONTACTS AND LOCATIONS:
Overall Officials: Shutian Zhang, MD, Principal Investigator — Beijing Friendship Hospital
Locations (18):
- China (18):
  - The Fourth Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital Affiliated to Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Shengjing Hospital Affiliated to China Medical University, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shandong Provincial Hospital, Jinan, Shandong
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Beijing Chaoyang Hospital Affiliated to Capital Medical University, Beijing
  - Beijing Friendship Hospital Affiliated to Capital Medical University, Beijing
  - Peking University Third Hospital, Beijing
  - Chongqing People's Hospital, Chongqing
  - Shanghai Oriental Hospital, Shanghai
  - Tianjin Medical University General Hospital, Tianjin